CLINICAL TRIAL: NCT01456286
Title: Randomized Trial, Masked, and Placebo Controlled to Assess the Effects of Sapropterin on Hepatic and Systemic Hemodynamics in Patients With Liver Cirrhosis and Portal Hypertension
Brief Title: Randomized Controlled Trial to Assess the Effects of Sapropterin on Hepatic and Systemic Hemodynamics in Patients With Liver Cirrhosis and Portal Hypertension
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Fundacion Clinic per a la Recerca Biomédica (Other)
Responsible Party: Principal Investigator, Sara Varea, Clinical Research Manager, Fundacion Clinic per a la Recerca Biomédica
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TEHYLIC
Record Dates: First submitted 2011-10-17; First posted 2011-10-20 (Estimated); Last update posted 2013-10-07 (Estimated); Status verified 2013-10

CONDITIONS: Liver Cirrhosis; Portal Hypertension
MeSH Terms: conditions — Liver Cirrhosis; Hypertension, Portal | interventions — sapropterin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sapropterin (Experimental): 5 mg/kg daily first week; 10 mg/kg daily second week of treatment
  Interventions: Drug: sapropterin
- placebo (Placebo Comparator)
  Interventions: Drug: sapropterin

INTERVENTIONS:
Drug: sapropterin — two weeks of treatment: 5 mg/kg per day during first week 10 mg/kg per day during second week

SUMMARY:
The purpose of this study is to determine whether sapropterin (an oral analogue of tetrahydrobiopterin) could have a role in the treatment of portal hypertension secondary to liver cirrhosis. Sapropterin or placebo will be given for two weeks in patients with liver cirrhosis and clinically significant portal hypertension. Systemic and hepatic hemodynamics studies will be performed at baseline and after the intervention to assess the effect of sapropterin.

DETAILED DESCRIPTION:
Portal hypertension and its complications (variceal bleeding, encephalopathy, spontaneous bacterial peritonitis, hepatorenal syndrome) are the main cause of death and liver transplantation in patients with cirrhosis. Diminishing portal hypertension by drugs (beta-blockers) is associated with a protection in the development of complications from portal hypertension. For this reason it is important to investigate and develop drugs that can reduce the portal pressure in liver cirrhosis. Tetrahydrobiopterin has been shown to decrease portal pressure in animal models of cirrhosis by improving intrahepatic resistance and by increasing nitric oxide bioavailability (eNOS co-factor). These effects were not associated to deleterious effects on systemic hemodynamics.

This study aims to test if sapropterin (an oral analogue of tetrahydrobiopterin) can play a role in the management of portal hypertension. For this, patients with liver cirrhosis and clinically significant portal hypertension will be randomized to receive sapropterin or placebo for two weeks. Patients will undergo an hepatic vein catheterization to asses the hepatic venous pressure gradient (HVPG), and those having and HVPG of 10 mmHg or higher will be randomized to receive sapropterin or placebo. Swan-Ganz catheterization, systemic measurements, and hepatic blood flow by indocyanine green method will also be performed. Patients will receive sapropterin or placebo for two weeks at a dosage of 5 mg/kg/d in the first week, increasing to 10 mg/kg/d in the second week if there are no adverse events or intolerance. A second systemic and hepatic hemodynamic study will be performed after 2 weeks of treatment to assess changes.

Changes in laboratory tests, liver function (Child-Pugh and MELD scores), endothelial dysfunction and oxidative stress markers (Von Willebrand Factor, Malondialdehyde) will be monitored during the study. As sapropterin has been never evaluated in cirrhotic patients, tolerance and adverse effects related to the medication will be registered.

The study will be stratified according to previous beta-blocker therapy (receiving or not receiving beta-blockers).

ELIGIBILITY:
Inclusion Criteria:

* Liver cirrhosis of any etiology diagnosed by biopsy or by clinical-imaging data
* Male or female patients between 18-75 years old in whom hepatic vein catheterization is indicated.
* Clinically significant portal hypertension defined by a HVPG ≥ 10 mmHg.
* Signed informed consent.

Exclusion Criteria:

* End-stage liver failure defined by one of the following: Prothrombin activity < 40% and/or Bilirubin > 5 mg/dl.
* Pregnancy or breastfeeding.
* Concomitant beginning of non-selective beta-blockers (propranolol, nadolol) during the administration of sapropterin. Beta-blockers are not exclusion criteria if they are on stable doses in the previous 6 weeks.
* Treatment with carvedilol or nitrates.
* Previous TIPS or derivative shunt.
* Hepatocellular carcinoma exceeding Milan criteria.
* Spontaneous bacterial peritonitis or any active infection when entering in the study.
* Portal vein thrombosis or cavernomatosis at ultrasound.
* Chronic heart failure, respiratory failure or chronic renal failure (Creatinine >2 mg/dl).
* Previous convulsions or epilepsy.
* Hypersensibility to sapropterin or any of its excipients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2011-10; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Changes in Hepatic Venous Pressure Gradient | 2 weeks
  Changes in portal pressure gradient as measured by hepatic vein catheterization, induced by 2 week treatment with sapropterin/placebo

CONTACTS AND LOCATIONS:
Overall Officials: Juan C García-Pagán, MD phD, Principal Investigator — Hospital Clínic of Barcelona
Locations (2):
- Spain (2):
  - Hospital Clínic de Barcelona, Barcelona, Barcelona
  - Hospital Ramón y Cajal, Madrid, Madrid Community